CLINICAL TRIAL: NCT07217236
Title: Evaluation of an Artificial Intelligence-Enhanced Electrocardiogram Strategy Versus Standard Care to Identify Patients Requiring Cardiac Implantable Electronic Devices: A Randomized Controlled Trial
Brief Title: Proactive Risk Evaluation for Cardiac Implantable Electronic Device Strategy Using AI-ECG
Acronym: PRECISE-AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Yu Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TSGH-AIECG-CIED
Record Dates: First submitted 2025-10-12; First posted 2025-10-15 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Artificial Intelligence (AI); Cardiac Implantable Electrical Devices; Conduction Disorder of the Heart
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AI-ECG prediction (Experimental)
  Interventions: Diagnostic Test: AI-ECG driven ECG monitoring
- Usual care (No Intervention)

INTERVENTIONS:
Diagnostic Test: AI-ECG driven ECG monitoring — Participants identified as high-risk for CIED implantation by the AI-ECG system will receive a continuous cardiac rhythm monitor for up to 7 days.
  Arms: AI-ECG prediction

SUMMARY:
The goal of this clinical trial is to learn whether an artificial intelligence-enhanced electrocardiogram (AI-ECG) strategy improves timely intervention of patients requiring cardiac implantable electronic devices (CIEDs), compared with standard clinical care.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to evaluate the impact of an AI-ECG strategy on the identification of patients requiring CIEDs. The ECGs of eligible participants will be analyzed by a previously validated deep learning algorithm. Those classified as high-risk by the AI-ECG system will be allocated at random into either the intervention group or the control group.

In the intervention group, the physicians will be alerted by the AI-ECG system, and the participants will be proactively contacted to receive ambulatory continuous ECG monitoring for up to 7 days. In the control group, the participants will continue with usual clinical care, and treating physicians will not have access to the AI-ECG results before the end of this study. To ensure accuracy, the reference standards for device indications will be performed by a panel of experienced cardiologists without access to the AI-generated reports.

ELIGIBILITY:
Inclusion Criteria:

* At least one 12-lead ECG within 1 year

Exclusion Criteria:

* Diagnosis of sick sinus syndrome
* Diagnosis of high-grade or complete atrioventricular block
* Diagnosis of ventricular tachycardia or ventricular fibrillation
* Post CIED implant
* Heart rate below 40 beats per minute by 12-lead ECG

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11492 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
CIED implantation | Within 180 days after randomization
  The number of participants who undergo CIED implantation within the study period. The CIEDs include conventional transvenous pacemakers, leadless pacemakers, and implantable cardioverter-defibrillators (encompassing transvenous, subcutaneous, and extravascular systems).

SECONDARY OUTCOMES:
Number of High-Grade Atrioventricular Block | Within 90 days after randomization
Number of Complete Atrioventricular Block | Within 90 days after randomization
Number of Sick Sinus Syndrome | Within 90 days after randomization
Number of Ventricular Arrhythmia | Within 90 days after randomization
Adverse Events Related to Continuous ECG Monitoring | Within 90 days after randomization.
  The number of adverse events associated with continuous ECG monitoring, including mild to moderate skin irritation, contact dermatitis, or discomfort at the site of patch application, as well as other procedure-related minor complications arising from extended ECG monitoring.
Number of CIED-Related Complications | Within 90 days after randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No